CLINICAL TRIAL: NCT03461692
Title: A Study of 100 Thousand Cases of Pediatric Patients of Clinical Safety Monitoring and Characteristic Observation and the Mechanism of Anaphylactic Reaction Used Reduning(a Chinese Medicine Injection)in Hospitals in China
Brief Title: A Registry Study of 100 Thousand Cases of Pediatric Patients on Reduning Injection（a Chinese Medicine Injection）Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Children's Hospital of Nanjing Medical University (Other); Hunan University of Traditional Chinese Medicine (Other); Qilu Children's Hospital of Shandong University (Other); Zhengzhou Children's Hospital, China (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RDN2018
Record Dates: First submitted 2018-02-11; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Upper Respiratory Tract Infection; Acute Tracheobronchitis
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Biospecimen Retention: Samples Without DNA — Under the patients'premise of consent and the signature of the informed consent, drawing the blood samples 5ml from the patients with allergic reactions and the patients without adverse reactions.The patients who responded to the 1:4 ratio matched the patients who had no adverse reactions (with the same sex, age difference within 5 years as the matching conditions）are intended for inflammatory factors to explore the mechanism of anaphylaxis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: patients under 14 years of age using Reduning injeciton — To assess in patients using Reduning injection's clinical features and drug adverse reaction during patients' hospital stay. The registry procedure will only for patients under 14 years of age using Reduning injection,observed from February 2018 to December 2018.

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in February 2018.

The purpose of this study is to make a monitoring of adverse reactions in 100 thousand children aged 14 years and below to see whether Reduning injection is safe and the characteristic and mechanism of anaphylactic reaction used Reduning injection in hospitals in China.

DETAILED DESCRIPTION:
In order to observe the clinical characteristics and adverse reactions of patients aged 14 and below using Reduning injection in hospital,registry study is suitable method in this area. Otherwise, nested case control study is used to find out the mechanism of anaphylaxis. Calculating the incidence of adverse drug reactions is one of the main aims for this study. 100000 cases need to be registered at least. The aim population is who using Reduning injection from February 2018 to December 2018.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 14 and below using Reduning injection from February 2018 to December 2018.

Exclusion Criteria:

None

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The aim population for observation of clinical characteristics and adverse reactionsis who using Reduning injection from February 2018 to December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Drug Reaction | 3 days
  Incidence of Reduning Injection'Adverse Drug Reaction（ADRs）and Identify Factors That Contributed to the Occurrence of the Adverse Drug Reaction

SECONDARY OUTCOMES:
The Ratio of Body Temperature to Normal | 3 days
  The Ratio of Body Temperature to Normal(Lower Than 37.3ºC)
The Ratio of WBC to Normal | 3 days
  The Ratio of Body Temperature to Normal(Within the Range of (4 to 10) x the 9 square of 10/L)
The Ratio of The Antibiotic Used | 3 days
  Calculating The Ratio of Patients Using Antibiotics Accounted for All Patients Using Reduning Injection.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No